CLINICAL TRIAL: NCT01907191
Title: Comparison of Bupivacaine to Liposomal Bupivacaine for Ultrasound Guided Periarticular Hip Infiltration for Postoperative Analgesia After Hip Arthroscopy.
Brief Title: Ultrasound Guided Local Infiltration Analgesia for Hip Arthroscopy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Trinity Health Of New England (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-06-001
Record Dates: First submitted 2013-06-28; First posted 2013-07-24 (Estimated); Results first posted 2022-07-19 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Hip Injuries
Keywords: Hip Arthroscopy; Liposomal Bupivacaine; Bupivacaine
MeSH Terms: conditions — Hip Injuries | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liposomal bupivacaine (Experimental): Ultrasound guided injection of liposomal bupivacaine for patients undergoing hip arthroscopy
  Interventions: Drug: liposomal bupivacaine
- Bupivacaine (Active Comparator): Bupivacaine (around the anterior, lateral and medial aspect of hip joint) for patients undergoing hip arthroscopy
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: liposomal bupivacaine — (Ultrasound guided injection of liposomal bupivacaine) for patients undergoing hip arthroscopy
  Other Names: Exparel
  Arms: Liposomal bupivacaine
Drug: Bupivacaine — (around the anterior, lateral and medial aspect of hip joint) for patients undergoing hip arthroscopy
  Other Names: Marcaine
  Arms: Bupivacaine

SUMMARY:
This study is being undertaken to compare the pain control using either bupivacaine versus liposomal bupivacaine. Liposomal bupivacaine can potentially provide pain relief lasting up to 72 hours while regular bupivacaine can provide pain relief up to 12 hours

DETAILED DESCRIPTION:
Patients undergoing hip arthroscopy experience moderate to severe postoperative pain. Effective pain control after surgery is an important component in the overall management of these patients. Good pain control encourages early participation in rehabilitation program, increases success of the surgery, and improves patient satisfaction. Typically, postoperative analgesia is provided to these patients either with nerve blocks or opioid medications. Both these methods provide good pain relief but nerve blocks are associated with weakness of lower extremity muscles which interferes with early ambulation and increase the risk of falls while narcotic medications increase the risk of nausea, vomiting, itching, constipation, ileus, urinary retention, sedation and respiratory depression.

ELIGIBILITY:
Inclusion Criteria:

* Patients having hip arthroscopy

Exclusion Criteria:

* History of neurologic disease, neuropathy, diabetes
* Allergy to local anesthetic solution
* Chronic use of narcotics
* Inability to give consent/cooperate with study
* History of previous hip arthroscopy on the ipsilateral side
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-07; Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Sinha, MD, Principal Investigator — Saint Francis Hospital and Medical Center
Locations (1):
- Saint Francis Hospital and Medical Center, Hartford, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Liposomal Bupivacaine: Ultrasound guided injection of liposomal bupivacaine
  liposomal bupivacaine: (Ultrasound guided injection of liposomal bupivacaine) for patients undergoing hip arthroscopy
- Bupivacaine: Bupivacaine (around the anterior, lateral and medial aspect of hip joint)
  Bupivacaine: (around the anterior, lateral and medial aspect of hip joint) for patients undergoing hip arthroscopy
Period: Overall Study
Arm/Group | Liposomal Bupivacaine | Bupivacaine
Started | 13 | 10
Completed | 13 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine | Liposomal Bupivacaine | Total
Number analyzed (Participants) | 10 | 13 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (8.9) | 30.5 (8.28) | 34.5 (10.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 6 | 6 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption (Mean Number of 5mg Oxycontin Tablets Consumed)
Description: Consumption of 5mg Oxycontin tablets will be assessed on Post Operative Days 1, 2 & 3.
Time Frame: Post Operative Day 1, 2 & 3
Measure: Mean (Standard Deviation); unit: number of 5 mg oxycontin
Arm/Group | Bupivacaine | Liposomal Bupivacaine
Number analyzed (Participants) | 10 | 13
number of 5 mg oxycontin
  Post Operative Day 1 | 2.8 (1.87) | 1.9 (1.50)
  Post Operative Day 2 | 2.7 (2.00) | 2.2 (2.34)
  Post Operative Day 3 | 2.3 (2.00) | 0.9 (1.38)

2. Secondary Outcome: Pain Scores
Description: Analysis of pain scores (at rest and ambulation) during hospital stay. Measured on a 10 point pain scale (1 being no pain and 10 being worst pain imaginable)
Time Frame: Post Operative Day 1, 2 & 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bupivacaine | Liposomal Bupivacaine
Number analyzed (Participants) | 10 | 13
score on a scale
  Pain Scores at rest- Post Operative Day 1 | 1.9 (0.94) | 1.1 (1.44)
  Pain Scores on Ambulation- Post Operative Day 1 | 3.1 (2.12) | 3.9 (2.43)
  Pain Scores at rest- Post Operative Day 2 | 1.9 (1.47) | 1.0 (1.35)
  Pain Scores on Ambulation- Post Operative Day 2 | 3.2 (1.0) | 3.1 (2.57)
  Pain Scores at rest- Post Operative Day 3 | 2.2 (1.87) | 1.6 (0.95)
  Pain Scores on Ambulation- Post Operative Day 3 | 2.6 (1.21) | 2.0 (1.44)

3. Other Pre Specified Outcome: Number of Patients Reporting Sleep Disturbance
Description: Analysis of sleep disturbance during hospital stay (participants who reported being woken up by pain on post operative days 1, 2 & 3)
Time Frame: Post Operative Day 1, 2 & 3
Measure: Count of Participants; unit: Participants
Arm/Group | Bupivacaine | Liposomal Bupivacaine
Number analyzed (Participants) | 10 | 13
Participants
  Post Operative Day 1 | 3 | 4
  Post Operative Day 2 | 3 | 3
  Post Operative Day 3 | 1 | 0

4. Other Pre Specified Outcome: Satisfaction With Pain Management
Description: Analysis of satisfaction with pain management during hospital stay measured on a 15 point scale (1 being extremely unsatisfied to 15 being extremely satisfied)
Time Frame: Post Operative Day 1, 2 & 3
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Bupivacine: Bupivacaine (around the anterior, lateral and medial aspect of hip joint) for patients undergoing hip arthroscopy
Arm/Group | Bupivacine | Liposomal Bupivacaine
Number analyzed (Participants) | 10 | 13
score on a scale
  Post Operative Day 1 | 13.9 (1.91) | 13.3 (2.69)
  Post Operative Day 2 | 14.1 (1.73) | 13.8 (2.24)
  Post Operative Day 3 | 14.6 (0.97) | 14.0 (2.22)

ADVERSE EVENTS:
Time Frame: Adverse events were collected until post operative day 3
Groups:
- Liposomal Bupivacaine: Ultrasound guided injection of liposomal bupivacaine
  liposomal bupivacaine: (Ultrasound guided injection of liposomal bupivacaine)
- Bupivacaine: Bupivacaine (around the anterior, lateral and medial aspect of hip joint)
  Bupivacaine: (around the anterior, lateral and medial aspect of hip joint)
Arm/Group | Liposomal Bupivacaine | Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/10
Other Adverse Events (participants affected / at risk) | 0/13 | 0/10

LIMITATIONS AND CAVEATS:
Study was terminated early leading to limited number of study subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-06-11): https://cdn.clinicaltrials.gov/large-docs/91/NCT01907191/Prot_SAP_000.pdf